CLINICAL TRIAL: NCT03747458
Title: 16-Week Randomized Double-Blind Placebo Controlled Parallel-Group Multicenter Study Evaluating the Efficacy and Safety of OPN-375 186 μg Twice a Day in Adolescents With Bilateral Nasal Polyps Followed With 12-Week Open-Label Treatment Phase
Brief Title: OPN-375 Efficacy and Safety in Adolescents With Bilateral Nasal Polyps
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPN-FLU-NP-3103
Record Dates: First submitted 2018-10-23; First posted 2018-11-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Bilateral Nasal Polyposis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OPN-375 186 μg BID (Active Comparator): Double-Blind Treatment Phase: OPN-375 186 μg BID x 16 weeks
  Open-Label Extension Phase: OPN-375 186 μg BID x 12 weeks
  Interventions: Drug: OPN-375
- Placebo (Placebo Comparator): Double-Blind Treatment Phase: Matching Placebo BID x 16 weeks
  Interventions: Drug: OPN-375

INTERVENTIONS:
Drug: OPN-375 — OPN-375, BID

SUMMARY:
This is a 16-Week Randomized, Double-Blind, Placebo Controlled, Parallel-Group, Multicenter Study Evaluating the Efficacy and Safety of OPN-375 186 μg Twice a Day (BID) in Adolescents with Bilateral Nasal Polyps followed by a 12-Week Open-Label Treatment Phase. The total planned number of subjects is approximately 72 adolescents (12-17 years of age) who will be randomly assigned to receive 1 of 2 study treatments using a 2:1 ratio (OPN-375 186 μg: Placebo). For the PK sub-study, up to 14 subjects will be enrolled to obtain 10 completers.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of intranasal administration of OPN-375 186 μg Twice a Day (BID) versus placebo in adolescents with bilateral nasal polyposis and nasal congestion by analyzing the reduction of nasal congestion/obstruction symptoms at the end of Week 4 measured by the 7-day average instantaneous morning diary symptom scores and the reduction in total polyp grade at Week 16 as determined by a nasal polyp grading scale score measured using a 0 to 6 point severity grading scale.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 12 to 17 years, inclusive, at time of Visit 1 (Screening).
2. Female subjects, if sexually active, must,

   1. be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [e.g., condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
   2. be surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or
   3. be abstinent.
3. All female subjects not documented to be infertile (e.g., infertility due to congenital abnormality or surgical sterilization) must have a negative serum or urine beta-human chorionic gonadotropin (hCG) at Visit 1 (Screening) and a negative urine pregnancy test at the Visit 2 (Day 1/Randomization/Baseline).
4. Must have bilateral nasal polyposis with a grade of 1 to 3 in each of the nasal cavities as determined by a nasal polyp grading scale score measured by nasoendoscopy at Visit 1 (Screening).
5. Must report at least mild symptoms of nasal congestion/obstruction as demonstrated by an average morning nasal congestion/obstruction score of at least 1.0 over a 7 day period during the single-blind run-in period. (Subjects not meeting this inclusion criterion may be re-screened once after at least 4 weeks.)
6. Subjects with comorbid asthma must be stable, defined as no exacerbations (e.g., no emergency room visits, hospitalization, or oral or parenteral steroid use) within the 3 months before Visit 1 (Screening). Subjects who received inhaled corticosteroids are required to be on no more than a moderate dosage regimen as defined by 2015 Global Initiative for Asthma Guidelines (GINA) for 1 month before Visit 1 (Screening) and to be expected to remain on it throughout the study (GINA 2015). Subjects receiving inhaled fluticasone alone or in combination may not participate in the PK sub-study.
7. Must be able to cease treatment with intranasal medications including, but not limited to, intranasal oxymetazoline or any other decongestants, intranasal antihistamines, intranasal steroids, intranasal sodium cromolyn, nasal atropine, nasal ipratropium bromide, inhaled corticosteroids (except permitted doses listed above for asthma) at Visit 1 (Screening). [Note: intranasal antibiotics and saline are permissible]
8. If taking oral antihistamines, must be on a stable regimen for at least 2 weeks prior to Visit 1 (Screening), and agree to not change the dose of these medications until after Visit 3 (Week 4) of the study.
9. Subjects (with assistance from parent or legal guardian if needed) must demonstrate the ability to complete the daily diary during the run-in period to be eligible for randomization.
10. Must demonstrate correct use of the demo EDS.
11. Must be capable, in the opinion of the investigator, of providing assent and the appropriate parent(s) or guardian must provide an informed consent to participate in the study.

Exclusion Criteria:

1. Pregnancy or lactation
2. Has a history of cystic fibrosis
3. Have used XHANCE (fluticasone propionate) nasal spray within the past 2 months
4. Inability to achieve bilateral nasal airflow for any reason, including nasal septum deviation
5. Inability to examine both nasal cavities for any reason, including severe nasal septum deviation
6. Have known history of nasal septum erosion, ulceration or perforation, or evidence of such lesion on Visit 1 (Screening) nasal examination/nasoendoscopy
7. Other significant nasal pathology or abnormal anatomy
8. Has had any episode of epistaxis with frank bleeding in the 3 months before Visit 1 (Screening)
9. History of more than 5 sinus or nasal surgeries for either nasal polyps or nasal/sinus inflammation (lifetime)
10. Have had any surgery on the nasal septum
11. History of sinus or nasal surgery within 6 months before Visit 1 (Screening)
12. History of any surgical procedure that prevents the ability to accurately diagnose or grade polyps
13. Current, ongoing rhinitis medicamentosa (rebound rhinitis)
14. Have significant oral structural abnormalities (e.g., a cleft palate)
15. History of Churg-Strauss syndrome or dyskinetic ciliary syndromes
16. Purulent nasal infection (recent fever or symptoms of lethargy), acute sinusitis, or upper respiratory tract infection within 2 weeks before Visit 1 (Screening). Potential subjects presenting with one of these infections may be rescreened after 4 weeks.
17. Have an allergy, hypersensitivity, or contraindication to corticosteroids or steroids
18. Have a hypersensitivity to any excipients in the study drug
19. Exposure to any glucocorticoid treatment with potential for systemic effects (e.g., oral or parenteral steroids, high dose topical steroids) within 1 month before Visit 1 (Screening); except as noted in inclusion criteria for subjects with comorbid asthma
20. Have received mepolizumab (Nucala®), reslizumab (Cinquair®), dupilumab (Dupixent®), omalizumab (Xolair®), or benralizumab (Fasenra™) within 6 months of Visit 1
21. Have nasal or oral candidiasis
22. Have taken a potent CYP3A4-inhibitor within 14 days before Visit 1 (Screening)
23. Any serious or unstable concurrent disease, psychiatric disorder, or any significant concomitant medical condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study, or pose a specific risk to the subject due to study participation
24. History or current diagnosis of any form of glaucoma or ocular hypertension (i.e., >21 mm Hg)
25. History of intraocular pressure elevation on any form of steroid therapy
26. Current diagnosis of the presence (in either eye) of a cataract of Grade 1 or greater as defined on the Eye Examination Worksheet OR, less than a Grade 1 cataract with associated visual impairment
27. A recent (within 1 year of Visit 1 [Screening]) history of drug or alcohol abuse or dependence
28. Positive urine drug screen at screening visit for stimulants, opioids, or cocaine
29. Have participated in an investigational drug clinical trial within 30 days of Visit 1 (Screening)
30. Parents, guardian or caregivers of the subject who are employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in nasal congestion/obstruction symptoms (mild, moderate, severe) at the end of Week 4 | 4 Weeks
  Change in nasal congestion/obstruction symptoms at the end of Week 4 measured by the 7-day average instantaneous morning (AM) diary symptom scores (ADS7-IA). The nasal symptom scale is what is used to score the nasal congestion/obstruction score, which is recorded in the diary. Nasal symptom scale is graded on a scale of 0=no symptom, 1=mild symptom, 2=moderate symptom, 3=severe symptom.
Mean change from baseline at Week 16 in total polyp grade | 16 Weeks
  Change in total polyp grade (sum of scores from both nasal cavities) at Week 16 as determined by a nasal polyp grading scale score measured using a 0 to 6 point severity grading scale, with 0 (no polyps) to 3 (severe polyps) points per nostril

SECONDARY OUTCOMES:
Change in bilateral polyp grade over time | 16 Weeks
  nasal polyp grading scale score measured using a 0 to 6 point severity grading scale, with 0 (no polyps) to 3 (severe polyps) points per nostril
Percentage of subjects with a ≥1 point improvement in polyp grade | 16 Weeks
  nasal polyp grading scale score measured using a 0 to 6 point severity grading scale, with 0 (no polyps) to 3 (severe polyps) points per nostril
Percentage of subject with a grade of 0 on at least one side of the nose | 16 Weeks
  nasal polyp grading scale score measured using a 0 to 6 point severity grading scale, with 0 (no polyps) to 3 (severe polyps) points per nostril
Change in diary symptom scores for the symptoms of nasal congestion/obstruction, measured as instantaneous and reflective scores for the morning and the afternoon (AM and PM scores) | 16 Weeks
  The Nasal Symptom Scale is graded on a scale of 0 (no symptom) to 3 (Severe symptom)
Change in diary symptom scores for the symptoms of rhinorrhea, measured as instantaneous and reflective scores for the morning and the afternoon (AM and PM scores) | 16 Weeks
  The Nasal Symptom Scale is graded on a scale of 0 (no symptom) to 3 (Severe symptom)
Change in diary symptom scores for the symptoms of facial pain or pressure, measured as instantaneous and reflective scores for the morning and the afternoon (AM and PM scores) | 16 Weeks
  The Nasal Symptom Scale is graded on a scale of 0 (no symptom) to 3 (Severe symptom)
Change in diary symptom scores for the sense of smell, measured as instantaneous and reflective scores for the morning and the afternoon (AM and PM scores) | 16 Weeks
  Sense of smell will be scored on a scale from 0 (normal) to 3 (absent, no sense of smell)
The proportions of subjects who have reductions in the AM and PM, instantaneous and reflective, average nasal congestion/obstruction symptom scores by 0.5 or more points from baseline to the end of the double-blind treatment phase | 16 Weeks
  The Nasal Symptom Scale is graded on a scale of 0 (no symptom) to 3 (Severe symptom)
Subjects will assess their global impression of change since starting the study drug using the PGIC scale | 16 Weeks
  Subject global impression of change will be assessed using a subject-completed PGIC scale, with a single question rated from 1=very much improved to 7=very much worse
Subjects will assess their change in quality of life since starting the study drug using the quality of life questionnaire (SN-5). | 16 Weeks
  Quality of life assessment using the SN-5 Questionnaire, a subject/parent-completed questionnaire that consists of 5 specific symptoms-related questions (answered on a 7-point Likert scale on the frequency of symptoms, 1=none of the time, 7=all of the time), and 1 general overall quality of life question (answered on a visual analog scale from 0 to 10, worst to best).
Proportion of subjects eligible for surgical intervention (independent of actual surgery performed) | Visit 1 (Screening) and Visit 6 (Week 16/ End of Double-Blind/Early Termination)
  The assessment criteria are as follows:
  * Subject has had moderate symptoms of congestion from nasal polyposis for at least 3 months.
  * Subject continues to suffer from at least moderate symptoms despite use of topical steroids at conventional doses for at least 6 weeks.
  * Subject continues to suffer from at least moderate symptoms despite use (or previous use) of saline lavage for at least 6 weeks.
  * Subject has endoscopically visualized bilateral nasal polyposis of at least moderate severity (nasal polyp grading score > 2 in at least 1 nostril). Also assess each subject's eligibility for surgery based on specific of criteria (see Section 12) independent of whether the subject actually undergoes surgery.

OTHER OUTCOMES:
Assessment of safety from physical examination-measuring weight | Visit 1 (Screening) and Visit 6 (Week 16/ End of Double-Blind/Early Termination)
  Assessment of safety from physical examination-weight measured in kg or lb
Assessment of safety from physical examination-measuring height | Visit 1 (Screening) and Visit 6 (Week 16/ End of Double-Blind/Early Termination)
  Assessment of safety from physical examination-height measured in cm or in
Assessment of safety by recording the severity of AEs | 16 Weeks
  Assessment of safety by measuring severity of AEs using scale with 1=mild, 2=moderate, 3=severe
Assessment of safety by nasal examination | 16 Weeks
  Assessed in nasal examination worksheet which includes recording the presence of any epistaxis, septal erosion/perforation, ulceration/erosion of area other than septum. If present, the nostril location is also recorded, along with severity, and if there is any relation to an injury or trauma
Assessment of safety by ocular examination-visual acuity | Visit 1 (Screening) and Visit 6 (Week 16/ End of Double-Blind/Early Termination)
  Assessment of safety by performing visual acuity test assessment using eye chart. Separate recording for each eye in the form of a fraction, 20/...
Assessment of safety by ocular examination-Intraocular Pressure | Visit 1 (Screening) and Visit 6 (Week 16/ End of Double-Blind/Early Termination)
  Assessment of safety by averaging intraocular pressure measurement of 2 or 3 measurements to determine if it is >21mmHg
Assessment of safety by ocular examination-Cataract Evaluation | Visit 1 (Screening) and Visit 6 (Week 16/ End of Double-Blind/Early Termination)
  Cataracts should be again assessed present or absent, If cataract is diagnosed, cataract type per localization should be specified and cataract should be graded 1=mild, 2=moderate, 3=pronounced, 4=severe
Assessment of safety measuring vital signs (blood pressure) | 16 Weeks
  Includes systolic and diastolic blood pressure measurements in millimeter of mercury (mmHg)
Assessment of safety measuring vital signs (pulse) | 16 Weeks
  measure pulse in beats per minute (bpm)
Assessment for safety from the collection of information for concomitant medications usage | 16 Weeks
Assessment of pharmacokinetics - AUC(0-t) (pg*hr/mL) | 8 hours, 1 to 2 weeks before randomization
  PK Laboratory to determine the concentrations of fluticasone propionate [AUC(0-t) (pg*hr/mL) measurement] in human plasma using high performance liquid chromatography (HPLC) with mass spectrometric detection. Approximately 5 mL of blood is collected from each subject at 10 different timepoints over an 8-hour period, for a total of 50 mL. The timepoints are: Pre-dose; 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 3 hours, 6 hours and 8 hours post-dose.
Assessment of pharmacokinetics - AUC(0-∞) (pg*hr/mL) | 8 hours, 1 to 2 weeks before randomization
  PK Laboratory to determine the concentrations of fluticasone propionate [AUC(0-∞) (pg*hr/mL) measurement] in human plasma using high performance liquid chromatography (HPLC) with mass spectrometric detection. Approximately 5 mL of blood is collected from each subject at 10 different timepoints over an 8-hour period, for a total of 50 mL. The timepoints are: Pre-dose; 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 3 hours, 6 hours and 8 hours post-dose.
Assessment of pharmacokinetics - AUCex (%) | 8 hours, 1 to 2 weeks before randomization
  PK Laboratory to determine the concentrations of fluticasone propionate [AUCex (%) measurement] in human plasma using high performance liquid chromatography (HPLC) with mass spectrometric detection. Approximately 5 mL of blood is collected from each subject at 10 different timepoints over an 8-hour period, for a total of 50 mL. The timepoints are: Pre-dose; 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 3 hours, 6 hours and 8 hours post-dose.
Assessment of pharmacokinetics - Cmax (pg/mL) | 8 hours, 1 to 2 weeks before randomization
  PK Laboratory to determine the concentrations of fluticasone propionate [Cmax (pg/mL) measurement] in human plasma using high performance liquid chromatography (HPLC) with mass spectrometric detection. Approximately 5 mL of blood is collected from each subject at 10 different timepoints over an 8-hour period, for a total of 50 mL. The timepoints are: Pre-dose; 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 3 hours, 6 hours and 8 hours post-dose.
Assessment of pharmacokinetics - tmax (h) | 8 hours, 1 to 2 weeks before randomization
  PK Laboratory to determine the concentrations of fluticasone propionate [tmax (h) measurement] in human plasma using high performance liquid chromatography (HPLC) with mass spectrometric detection. Approximately 5 mL of blood is collected from each subject at 10 different timepoints over an 8-hour period, for a total of 50 mL. The timepoints are: Pre-dose; 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 3 hours, 6 hours and 8 hours post-dose.
Assessment of pharmacokinetics - t1/2 (h) | 8 hours, 1 to 2 weeks before randomization
  PK Laboratory to determine the concentrations of fluticasone propionate [t1/2 (h) measurement] in human plasma using high performance liquid chromatography (HPLC) with mass spectrometric detection. Approximately 5 mL of blood is collected from each subject at 10 different timepoints over an 8-hour period, for a total of 50 mL. The timepoints are: Pre-dose; 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 3 hours, 6 hours and 8 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Manley, Study Chair — Paratek Pharma
Locations (40):
- United States (31):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - San Tan Allergy & Asthma, Gilbert, Arizona
  - Kern Research, Bakersfield, California
  - Central California Clinical Research, Fresno, California
  - Sensa Health, Los Angeles, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Allergy and Asthma Consultants, Redwood City, California
  - Sacramento ENT, Roseville, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale School of Medicine, Section of Otolaryngology, New Haven, Connecticut
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush University Medical Center - Department of Otorhinolaryngology, Chicago, Illinois
  - Chicago ENT, Chicago, Illinois
  - Kentuckiana ENT, Louisville, Kentucky
  - Ochsner Medical Center, Otorhinolaryngology Department, New Orleans, Louisiana
  - Children's Minnesota, Minneapolis, Minnesota
  - University of Missouri Medical Center, Columbia, Missouri
  - University of Rochester, Rochester, New York
  - Allergy Asthma & Immunology Research Institute, Charlotte, North Carolina
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - MUSC Department of Otolaryngology, Head and Neck Surgery, Charleston, South Carolina
  - Carolina ENT, Orangeburg, South Carolina
  - STAAMP Research, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School - Otolaryngology, Norfolk, Virginia
  - Spokane ENT, Spokane Valley, Washington
  - West Virginia University, Morgantown, West Virginia
- Argentina (9):
  - Instituto Medico Rio Cuarto, Río Cuarto, Córdoba Province
  - Instituto Medico de la Fundacion de Estudios Clinicos - Consultorios Integrados Rosario, Rosario, Santa Fe Province
  - Centro de Investigaciones Clinicas - Instituto de la Salud Rosario, Rosario, Santa Fe Province
  - Clinica Mayo, UMCB, San Miguel de Tucumán, Tucumán Province
  - Sanatorio Guemes, Buenos Aires
  - Fundacion CIDEA, Buenos Aires
  - InAER - Investigaciones en Alergia y Enfermedades Respiratorias, Buenos Aires
  - Instituto de Asma Alergia y Enfermedades Respiratoria (IAAER), Corrientes
  - Centro Medico INSARES, Mendoza